CLINICAL TRIAL: NCT00321269
Title: Depression and CHF in Outpatients
Brief Title: Depression and Congestive Heart Failure in Outpatients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: IIR 06-082
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure; Depression
Keywords: Home Monitoring; Heart Failure; Depression
MeSH Terms: conditions — Heart Failure; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Illness Managment (Active Comparator): This intervention includes standard disease self-management coaching for heart failure and helps patients set goals for fluid management, restricted salt-intake, and medication adherence.
  Interventions: Behavioral: Single Illness Management
- Comorbid Illness Management (Experimental): This intervention includes the same self-management coaching found in the comparator arm, but also includes discussion of ways to cope and manage mood.
  Interventions: Behavioral: Comorbid Illness Management

INTERVENTIONS:
Behavioral: Single Illness Management — 8 week nursing intervention addressing Congestive Heart Failure
  Arms: Single Illness Managment
Behavioral: Comorbid Illness Management — 8 week nursing intervention to address Congestive Heart Failure and emotional coping
  Arms: Comorbid Illness Management

SUMMARY:
Patients with a diagnosis of CHF, NYHA class II, III or IV will be recruited for a study comparing a nursing intervention addressing CHF (SIM group) or CHF and depression (CIM group). Participants in the standard illness management program will receive an 8-week, 8-session intervention designed to help them improve daily weighing, salt-restriction, medication management, etc. This intervention will be conducted in a combination of home visits and phone visits. They will also receive interactive, telephone-based daily monitoring that assesses daily weight, dyspnea, fatigue and medication compliance. Patients in the comorbid illness management program will receive the same illness management program PLUS education and behavioral techniques designed to help them cope emotionally with the illness. The comorbid illness management home monitoring will include a twice-monthly screen for depression. Major Variables: The major outcomes will be depressive symptoms, health-related quality of life, functional status, heart failure symptom severity, and self-care behaviors in heart failure.

DETAILED DESCRIPTION:
Background:

Between 4 and 5% of patients seen at Veterans Affairs Medical Centers suffer heart failure. HF is the number one discharge diagnosis within the VHA. One of the most significant comorbidities in heart failure is depression. Depression predicts increased hospitalization and mortality even after controlling for key prognostic indicators. This HSR&D study aimed to test the effectiveness of a psychotherapy intervention for depression combined with illness management to illness management alone in veterans with heart failure.

Objectives:

To demonstrate better depression, health-related quality-of-life, and adherence outcomes for an illness management combined with psychotherapy intervention (COMBO) as compared to an illness management alone program (IMO).

Methods:

This was a two-site, two-arm, randomized controlled trial comparing COMBO to IMO. The total number of patients recruited for the study was 148. Retention was comparable between groups, though depression severity predicted drop out in the IMO condition but not the COMBO condition. Patients completed study assessments at baseline, week 4, week 8 (post-intervention) and at 26- and 52-week follow-up.

Status:

The main study analyses have been conducted. The project team is conducting analysis of secondary hypotheses

ELIGIBILITY:
Inclusion Criteria:

* Receiving treatment for NYHA Class 2-4 heart failure.
* Patients of the Iowa City, IA or Columbia, MO Veterans Affairs Medical Center Primary Care or Cardiac Care Clinics.
* Life expectancy greater than 6 months.
* Must speak English.
* Must possess a working telephone.

Exclusion Criteria:

* Presence of major psychiatric illness such as schizophrenia, bipolar disorder and substance abuse (PTSD patients are eligible).
* Life expectancy less than 3 months.
* Planned relocation to a nursing home.
* Marked visual or hearing impairment.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn L Turvey, PhD MS, Principal Investigator — VA Medical Center, Iowa City
Locations (2):
- United States (2):
  - Iowa City VA Medical Center, Iowa City, Iowa
  - Harry S. Truman Memorial VA Medical Center, Columbia, Missouri

REFERENCES:
- [Result] Turvey C, Sheeran T, Dindo L, Wakefield B, Klein D. Validity of the Patient Health Questionnaire, PHQ-9, administered through interactive-voice-response technology. J Telemed Telecare. 2012 Sep;18(6):348-51. doi: 10.1258/jtt.2012.120220. Epub 2012 Aug 29. PMID 22933480

RESULTS

PARTICIPANT FLOW:
Groups:
- 8-week Phone Based Single Illness Management: Standard nursing intervention to treat Congestive Heart Failure
  Education & behavioral techniques to help CHF patients cope with chronic illness: 8 week nursing intervention addressing Congestive Heart Failure
- 8-week Phone Based Comorbid Illness Management: Nursing intervention to treat Congestive Heart Failure and emotional coping
  CHF and emotional coping: 8 week nursing intervention to address Congestive Heart Failure and emotional coping
Period: Overall Study
Arm/Group | 8-week Phone Based Single Illness Management | 8-week Phone Based Comorbid Illness Management
Started | 74 | 74
Completed | 66 | 68
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- 8-Week Phone-based Comorbid Illness Management: Nursing intervention to treat Congestive Heart Failure and emotional coping
  CHF and emotional coping: 8 week nursing intervention to address Congestive Heart Failure and emotional coping
- Total: Total of all reporting groups
Arm/Group | 8-week Phone Based Single Illness Management | 8-Week Phone-based Comorbid Illness Management | Total
Number analyzed (Participants) | 66 | 68 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (8.9) | 67.8 (9.1) | 70.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 65 | 66 | 131
Region of Enrollment [Number; unit: participants]
  United States | 66 | 68 | 134

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory II
Description: Depressive Symptoms measured on a Beck Depression Inventory Revised Possible Range 0 to 63. Higher scores indicate greater depression. Effectiveness of treatment indicated by a decline in the BDI-II score.
Time Frame: Depression and psychological health will be assessed at week 1, week 8
Population: Older Veterans with Heart Failure
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 8-week Phone-based Single Illness Management: Standard nursing intervention to treat Congestive Heart Failure
  Education & behavioral techniques to help CHF patients cope with chronic illness: 8 week nursing intervention addressing Congestive Heart Failure
Arm/Group | 8-week Phone-based Single Illness Management | 8-week Phone-based Comorbid Illness Management
Number analyzed (Participants) | 66 | 68
units on a scale
  Week 1 | 9.3 (0.85) | 9.2 (0.84)
  Week 8 | 9.0 (0.95) | 8.6 (0.96)
Statistical Analysis 1: Comparison: 8-week Phone-based Single Illness Management vs 8-week Phone-based Comorbid Illness Management; Mixed effects regression analysis- Treatment Arm X Time F (2, 116)=0.09, P>F=0.90; Test type: Superiority or Other; p = 0.90, Mixed Models Analysis

2. Secondary Outcome: Health-Related Quality of Life
Description: Medical Outcomes Study SF-36 Physical Function Subscale- 10 Items Range 0 to 100, Higher Scores indicate higher functioning.
Time Frame: Measured at week 1, week 8
Population: Older Veterans with Congestive Heart Failure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Phone-Based Single Illness Management | 8-Week Phone-Based Comorbid Illness Management
Number analyzed (Participants) | 66 | 68
units on a scale
  Week 1 | 36.82 (2.7) | 37.2 (2.7)
  Week 8 | 36.5 (2.9) | 43.1 (2.9)
Statistical Analysis 1: Comparison: 8-Week Phone-Based Single Illness Management vs 8-Week Phone-Based Comorbid Illness Management; Test type: Superiority or Other; p = 0.13, Mixed Models Analysis; F(2,110)=2.08; P=0.13

ADVERSE EVENTS:
Time Frame: 8 weeks- duration of the clinical trial. Adverse event was assessed at Week 4 and Week 8.
Description: Participants indicating depression were assessed for suicidality and any mortality due to suicide was monitored. These were the only adverse events monitored specifically.
  Suicidal ideation was assessed using the Beck Depression Inventory (Question #9) and the Structured Clinical Interview for DSM (Suicidal ideation question).
Groups:
- 8-week Telephone Based Single Illness Management: Standard nursing intervention to treat Congestive Heart Failure
  Education & behavioral techniques to help CHF patients cope with chronic illness: 8 week nursing intervention addressing Congestive Heart Failure
Arm/Group | 8-week Telephone Based Single Illness Management | 8-Week Phone Based Comorbid Illness Management
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/68
Other Adverse Events (participants affected / at risk) | 0/66 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8-week Telephone Based Single Illness Management (N=66) | 8-Week Phone Based Comorbid Illness Management (N=68)
Suicide (Psychiatric disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No